CLINICAL TRIAL: NCT01189708
Title: Prevention of Incisional Hernia After Elective Open Abdominal Aortic Aneurysm Repair
Brief Title: Prevention of Incisional Hernia After Elective Open Abdominal Aortic Aneurysm (AAA) Repair
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Treatment without success, low enrollment, one serious adverse event
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Ignazio Tarantino, M.D., Cantonal Hospital of St. Gallen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EKSG08/006
Record Dates: First submitted 2008-02-20; First posted 2010-08-27 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal aortic aneurysm; Abdominal hernia
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Hernia, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mesh implantation (Experimental): Ultrapro® Mesh implantation
  Interventions: Device: Ultrapro® Mesh implantation
- Standard wound closure without a mesh (Active Comparator): Standard wound closure
  Interventions: Other: Standard wound closure

INTERVENTIONS:
Device: Ultrapro® Mesh implantation — After the aortic procedure (aortic aneurysm repair) an Ultrapro absorbable mesh will be used for the wound closure of the abdominal wall using an onlay technique.
  Arms: Mesh implantation
Other: Standard wound closure — Abdominal closure will be performed with standard sutures without a mesh.
  Arms: Standard wound closure without a mesh

SUMMARY:
The aim of this study is to investigate the effect of the implantation of an Ultrapro® Mesh as prevention of incisional hernia after elective open abdominal aortic aneurysm repair. According to the literature these patients have an increased risk for an incisional hernia. By the implantation of an artificial mesh into the abdominal wall during the first abdominal aortic aneurysm repair, the risk can be reduced dramatically. In small feasibility studies incisional hernia rates as low as 0% have been achieved.

Patients scheduled for elective open abdominal aortic aneurysm repair will be randomized into two groups, one receiving an onlay mesh, the other conventional wound closure with sutures.

DETAILED DESCRIPTION:
Prospective randomized controlled study with two study arms.

Arm 1: Abdominal wall will be closed with a prophylactic mesh implantation in onlay technique after elective open abdominal aortic aneurysm repair.

Arm 2: Abdominal wall will be closed with standard sutures (without mesh implantation)

After the patients gave their informed consent to participate in the study, they will be randomized to one of the two treatment arms. Allocation is carried out based on a prepared randomization list.

Primary endpoint is the rate of incisional hernias within the follow-up period of 2 years. Secondary endpoints are postoperative complications and adverse events during the follow-up period.

Study enrollment was prematurely terminated on 30. Apr 2009. Already enrolled patients will be followed for 24 months according to protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for elective or early elective open repair of aortic aneurysm

Exclusion Criteria:

* Emergency surgery
* EVAR (endovascular procedure)
* Patients with previous midline laparotomy
* Patients with in situ abdominal mesh after previous hernia repair
* Patients with large diastasis of abdominal wall
* Allergy to penicillin
* Women before menopause (mesh can interfere with potential future pregnancies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Incidence of incisional hernia | 24 months

SECONDARY OUTCOMES:
Rate of postoperative complications | 7 days
operation time | 4 hours
Rate of adverse events | 24 months
  Adverse events related to mesh implantation

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Nagel, MD, Principal Investigator — KSSG
Locations (1):
- Kantonsspital St. Gallen, Department of Surgery, Sankt Gallen, Canton of St. Gallen, Switzerland